CLINICAL TRIAL: NCT03421587
Title: Abnormal Processing of Stressful Social Stimuli After Trauma Exposure, in Particular After Childhood Maltreatment.
Brief Title: Perception of Stressful Social Stimuli After Trauma Exposure.
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Vice Chair of the Department of Psychiatry and Chair of the Medical Psychology Division, University Hospital, Bonn
Other Study IDs: TT-Study
Record Dates: First submitted 2016-08-12; First posted 2018-02-05 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Individuals exposed to an intentional/non-intentional trauma
  Interventions: Behavioral: Processing of social olfactory and tactile stimuli
- Healthy controls without trauma-exposure
  Interventions: Behavioral: Processing of social olfactory and tactile stimuli

INTERVENTIONS:
Behavioral: Processing of social olfactory and tactile stimuli — Processing of social olfactory and tactile stimuli in trauma-exposed individuals and controls is examined using functional magnetic resonance imaging.

SUMMARY:
Post-traumatic stress disorder is associated with altered processing of sensory stimuli. The clinical phenotype PTSD has predominantly been described for the visual and auditory sensory modalities. However, PTSD symptoms such as intrusive memories are often evoked by olfactory and tactile cues in the environment. Moreover, little is known about whether aberrant responses to social olfactory and tactile stimuli are also present in a subclinical population.The purpose of this study is to compare trauma-exposed subjects (e.g. childhood maltreatment) with non-exposed controls in the processing of olfactory and tactile stimuli. This sensory characterizations hold potential to identify potential biomarkers for the course of trauma-related disorders and to inform trauma therapies focusing on sensory integration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects that have experienced a traumatic event that meets the DSM-5 criteria

Exclusion Criteria:

* Schizophrenia, schizoaffective or other psychotic disorder
* Neurological disorders
* Psychotropic medication
* Subjects suffering from a respiratory tract infection or other respiratory disorder known to affect olfactory functioning at investigator's discretion
* Subjects with anosmia or other previous primary olfactory dysfunction (olfactory threshold score using the "Sniffin' Sticks" ≤ 5)
* Dermatitis of the extremities or other skin disorders that affect the skin sensitivity of the extremities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of trauma-exposed subjects and healthy controls without trauma-exposure.Patients and healthy controls will be recruited from the Bonn area.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Emotion recognition ratings obtained during a forced-choice emotional face recognition task with stimuli of varying intensities (neutral to fearful). | Ratings will be assessed throughout fMRI scanning over the course of 25 minutes.
Neural substrates of social tactile stimuli processing. | The neural substrates will be assessed througout fMRI scanning over the course of 20 minutes.
  fMRI scanning will be used to measure neural respones to tactile stimuli.
Valence ratings of social tactile stimuli. | Ratings will be assessed throughout fMRI scanning over the course of 20 minutes.
Neural substrates of social olfactory stimuli processing. | The neural substrates will be assessed througout fMRI scanning over the course of 25 minutes.

SECONDARY OUTCOMES:
Oxytocin plasma concentrations. | The oxytocin plasma concentrations of all participants will be assessed 15 minutes before fMRI scanning onset..
Olfactory performance in a n-butanol odor staircase threshold test. | The olfactory threshold of all participants will be assessed in a screening session at least 24 hours prior to fMRI scanning.
  Participants' olfactory performance will be assessed by administering the 'Sniffin' Sticks' test, which measures nasal chemosensory performance based on pen-like odor dispensing devices.

CONTACTS AND LOCATIONS:
Overall Officials: René Hurlemann, PhD, MD, MSc, Principal Investigator — Department of Psychiatry, University of Bonn, Germany
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, Germany

REFERENCES:
- See also: Related Info — http://renehurlemann.squarespace.com/welcome/